CLINICAL TRIAL: NCT04157023
Title: Direct-Ophthalmoscopy-Simulator-Study
Brief Title: Simulator Training for Direct Ophthalmoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Dr. Martin Leitritz, Principle Investigator, University Hospital Tuebingen
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Simulator
Record Dates: First submitted 2019-11-01; First posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Simulator-based Medical Skill Training
Keywords: simulator; medical skills

STUDY DESIGN:
Intervention Model Description: Three groups of participants are made. Group 1: Medical Students Group 2: Ophthalmologists Group 3: Neonatologists/Neurologists/Neurosurgeons
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Medical Students (Other): Simulator training of 7 patient cases adapted to medical students.
  Interventions: Device: Simulator-based Training of Direct Ophthalmoscopy
- Ophthalmologist (Other): Simulator training of 7 patient cases adapted to ophthalmologists.
  Interventions: Device: Simulator-based Training of Direct Ophthalmoscopy
- Neurologist/Neurosurgeon/Neonatologist (Other): Simulator training of 7 patient cases adapted to neurologists, neurosurgeons and neonatologists.
  Interventions: Device: Simulator-based Training of Direct Ophthalmoscopy

INTERVENTIONS:
Device: Simulator-based Training of Direct Ophthalmoscopy — A digital simulator is used to teach the skills of direct ophthalmoscopy

SUMMARY:
Evaluation of a digital simulator to train diagnostic skills in Ophthalmology

DETAILED DESCRIPTION:
Direct Ophthalmoscopy is an important tool to detect pathologies e.g. on the optic nerve head. The training of the needed skills is made conventionally in most cases. In such the training sessions students examine each other after dilating one pupil. Examining of patients with pathologies is very important, but in many cases not very easy without any experience.

Simulators are of growing impact to teach diagnostic or surgical skills. A digital simulator with virtual reality technology is used to teach the skills to unexperienced examiners. The head-eye-hand-coordination can be trained without any stress.

ELIGIBILITY:
Inclusion Criteria:

* Medical student or Ophthalmologist or Neonatologist or Neurologist or Neurosurgeon
* Willing to participate to the study
* Consent to evaluate the measured data

Exclusion Criteria:

* age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Total examined area | 1 hour
  The area that was examined (light on retina) by participants was measured [percent of total area].
Efficiency | 1 hour
  Ratio of examination time (light in pupil) and total examined area [ratio]

SECONDARY OUTCOMES:
Learning effect | 1 hour
  Total examined area results and efficiency ratios were compared between simulator case 1 and simulator case 5.
Questionnaire | 1 hour
  A questionnaire was used to measure the self-evaluation of the trained persons

IPD SHARING:
Plan to Share IPD: No